CLINICAL TRIAL: NCT03262298
Title: Anti-CD22 Chimeric Antigen Receptor (CAR)-Modified T Cell Therapy Targeting CD22 in Treating Patients With B Cell Malignancies
Brief Title: Anti-CD22 CAR-T Cell Therapy Targeting B Cell Malignancies
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 307-B-22-CAR-T
Record Dates: First submitted 2017-08-14; First posted 2017-08-25 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Leukemia; Lymphoma
Keywords: CD22; CAR-T; Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD22 CAR-T (Experimental): Patients will receive a full dose CART infusion at day 0.
  Interventions: Biological: Anti-CD22-CAR-transduced T cells

INTERVENTIONS:
Biological: Anti-CD22-CAR-transduced T cells — a single dose of Anti-CD22-CAR-transduced T cells will be infusion after preconditioning.
  Other Names: anti-CD22 CART, CART22

SUMMARY:
The study will evaluate safety and efficacy of the CD22-targeted chimeric antigen receptor modified-T cell(CAR-T) cells in the treatment of B-cell Malignancies.

DETAILED DESCRIPTION:
Clinical success with chimeric antigen receptor (CAR)- based immunotherapy for leukemia has been accompanied by the associated finding that antigen-escape variants of the disease are responsible for relapse. Despite anti-CD19 CAR-T exhibited the ability to re-induce remissions for many patients with relapsed and refractory B cell malignancies, a part of those patients will relapse with CD19-negative malignancies. CD22 is a type I transmembrane protein expressed on most mature B lymphocyte in the B cell malignancies，and plays a significant role in signal transduction pathway. The investigators design and conduct this trial to test the safety and effectiveness of CD22-targeted CAR-T.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 years
2. Patients with Cluster of Differentiation 22(CD22) positive B cell malignancies as confirmed by flow cytometry
3. Refractory or relapsed B cell-acute lymphoblastic leukemia
4. No available curative treatment options (such as hematopoietic stem cell transplantation)
5. Stage III-IV disease
6. Creatinine < 2.5 mg/dl
7. Aspartate transaminase-alanine transaminase ratio < 3x normal
8. Bilirubin < 2.0 mg/dl
9. Karnofsky performance status >= 60
10. Expected survival time > 3 months
11. Adequate venous access for apheresis
12. Ability to understand and provide informed consent

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients requiring T cell immunosuppressive therapy
3. Active central nervous system leukemia
4. Any concurrent active malignancies
5. Patients with a history of a seizure disorder or cardiac disorder
6. Previous treatment with any immunotherapy products
7. Patients with human immunodeficiency virus, hepatitis B or C infection
8. Uncontrolled active infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2022-08-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events related to treatment as assessed by NCI CTCAE version 4.03 | 2 years

SECONDARY OUTCOMES:
Overall Complete Remission Rate (ORR) | 2 years
Disease response(CR, CRi) | 2 years
CART cells persistence in vivo | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Liangding Chen, M.D., Principal Investigator — Affiliated Hospital to Academy of Military Medical Sciences
Locations (1):
- Fengtai District, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided